CLINICAL TRIAL: NCT06404307
Title: Self-administration in Outpatient Parenteral Antimicriobial Therapy Service
Brief Title: Self-administration in Outpatient Parenteral Antimicrobial Therapy Service
Acronym: SELF-OPAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Amphia Hospital (Other)
Responsible Party: Principal Investigator, Dr. B.C.M. (Brenda) de Winter, Assistent professor, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ABR NL85913.078.24
Record Dates: First submitted 2024-04-09; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Infections; Bacterial Infections
Keywords: Outpatient; Antimicrobials; Outpatient Parenteral Antimicrobial Treatment
MeSH Terms: conditions — Infections; Bacterial Infections | interventions — Self Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-administration (Experimental): Trained patients that will self-administer their antimicrobials in the outpatient setting
  Interventions: Behavioral: Self-administration

INTERVENTIONS:
Behavioral: Self-administration — patients will self administer their antimicrobial treatment

SUMMARY:
Home Outpatient Parenteral Antimicrobial Treatment (Home-OPAT) is a service provided to patients that receive antibiotics via infusion but are clinically well enough to go home. A nurse will visit the patient daily to administer the antibiotics. However, the patient or a caregiver can also administer the antibiotics without the help of a nurse. This is called Self-OPAT. The Self-OPAT service is already in practice internationally but not yet in the Netherlands.

The goal of this observational study is to assess the possibility to implement Self-OPAT in the Dutch context. The main questions it aims to answer are:

Which patients are suitable for Self-OPAT services? How can patients be trained adequately for performing Self-OPAT? What are the experiences of patients with Self-OPAT? How much nurse engagement is needed during Self-OPAT? Is the outcome of treatment with Self-OPAT comparable to Home-OPAT? How do the costs of Self-OPAT differ from the costs of Home-OPAT? How can you implement an Self-OPAT program in the hospital?

Participants will be trained by a nurse to administer the infusion antibiotics. They will then administer the antibiotics themselves for as long as the duration of treatment. Every week a nurse will visit to check the progression of the treatment and check the functioning and hygiene of the infusion materials. After a month participants will fill-out a questionnaire about their experience with Self-OPAT.

DETAILED DESCRIPTION:
Outpatient parenteral antimicrobial therapy (OPAT) is defined as 'the administration of parenteral antimicrobial therapy in at least 2 doses on different days without intervening hospitalization. It can be provided for patients who need parenteral therapy for severe or deeply seated infections, under the condition that they are stable and healthy enough to leave the hospital. Nowadays, OPAT is considered regular care in many countries across Europe, Asia, North America, and Oceania. It is a safe, effective, and cost-saving practice.

OPAT can be performed in a variety of models. Infusion in the patient's home with active intervention of nursing personnel is called 'Healthcare Professional Outpatient Parenteral Antimicrobial Therapy (H-OPAT). In the Netherlands, the H-OPAT model is common practice. A disadvantage of H-OPAT is the need to arrange a nurse (from a home care organization) for visiting the patient at home to administer the intravenous antimicrobial.

Home-based H-OPAT can also be performed by the patient or a caregiver, introducing another model called self-administration OPAT (S-OPAT). In this model, healthcare personnel initially trains the patient and/or their caregivers to administer antimicrobials. After training, the patient or the caregiver administrates the intravenous antimicrobial instead of a visiting nurse. Internationally, S-OPAT is a well-established practice and it is known that it is a safe and effective practice and leads to increased patient satisfaction and reduced healthcare costs.

This is a prospective observational feasibility study to assess the feasibility of self-administration of intravenous antimicrobial therapy in the Dutch context.

Due to research lacking on S-OPAT in the Netherlands and the limited experience with S-OPAT in the Netherlands the following questions are still to be answered:

* Which patients are suitable for S-OPAT?
* How can patients be trained adequately for performing S-OPAT?
* What are the experiences of patients with S-OPAT?
* How much nurse engagement is needed during S-OPAT?
* Are the clinical outcomes with S-OPAT comparable to H-OPAT?
* What is the cost benefit of S-OPAT?
* How can you implement an S-OPAT program in the hospital?

After inclusion into the study the patient or a caregiver will be trained to perform S-OPAT by a nurse. The nurse will then sign a qualification form. If a patient is deemed unsuitable they will be deferred to the regular OPAT program. In the study there will be a weekly mandatory visit from the nurse of the home care organization for line dressing change and line care. The weekly home visits provide opportunities to assess patient condition and adherence to the self-administration. The patient's ongoing ability to perform self-administration and care partner fatigue are also evaluated. For this assessment, the nurse will fill out a short check-list every week. If during the S-OPAT trajectory, the patient is deemed unsuitable to perform self-administration according to the visiting nurse, the patient/caregiver will stop self-administration and will be deferred to the regular OPAT program. At day 30 after discharge, patients will be asked to fill out questionnaires regarding: health-related quality of life, acceptability and satisfaction with the S-OPAT service.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Hospitalized
* Treated with intravenous antimicrobial therapy and to be discharged with OPAT service
* To be discharged with OPAT service for a minimum of 5 days
* Central intravenous access/line in place
* Has a safe home environment (water, telephone, refrigerator available) and access to transport to hospital
* Able to understand written information and able to give informed consent
* Able and willing to perform self-administration, or able and willing to be self-administered by family members or other caregivers
* Able and willing to fill in questionnaires

Exclusion Criteria:

* Former participation in this study
* Pregnancy
* Discharge to a rehabilitation centre or nursing care centre (i.e. no discharge to home)
* Concomitant nursing care, if the patient requires other nursing care the patient will be placed on nursing care and the nurses administer the medication during the concomitant nursing care
* More than two intravenous drugs required
* More than one intravenous administration device required (e.g. elastomeric pump and medication cassette)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
To asses the capability of patients to self-administer antibiotics in the outpatient setting in the Dutch medical system. | 30 days after discharge
  To assess the feasibility of self-administration of intravenous antimicrobial therapy in the Dutch context. Feasibility is defined as adherence to the study protocol, which is defined as qualification for S-OPAT after training and completing an S-OPAT trajectory with a weekly scheduled nurse visit.

SECONDARY OUTCOMES:
Visits | 30 days after discharge
  To investigate the number of scheduled and unscheduled S-OPAT related nurse visits to the patient
Consultations | 30 days after discharge
  To investigate the number of OPAT related telephone consultations (to the nurse and the hospital)
Devices | 30 days after discharge
  To investigate the number of the different infusion devices (i.e. elastomeric pumps, infusion bags, infusion cassettes) used for S-OPAT patients in this study
Time to discharge | 30 days after discharge
  To investigate the time to discharge after signing up for OPAT
Training completion | 30 days after discharge
  The number of patients/caregivers who successfully complete S-OPAT training and are therefore qualified for self-administration.
Patient/caregiver characteristics | 30 days after discharge
  To describe characteristics of patients/caregivers who successfully completed S-OPAT training versus patients who did not qualify for self-administration.
  To describe characteristics of patients/caregivers who successfully completed their S-OPAT trajectory (with only a weekly scheduled nurse visit) versus patients who did not.
The number of patients/caregivers who finish their complete assigned S-OPAT trajectory | 30 days after discharge
  The total amount of patients or caregivers that succesfully complete their assigned S-OPAT trajectory.
The costs associated with performing and organizing S-OPAT in de Dutch medical system | 30 days after discharge
  To investigate the healthcare costs of S-OPAT by investigating the costs attributed to:
  * loss of productive hours by the patient
  * requirement of nursing staff
  * travel costs
  * cost of materials
Clinical outcomes: The outcomes of the infection in S-OPAT treatment | 30 days after discharge
  To investigate the progression of the infection in the patients when in S-OPAT treatment.
Clinical outcomes: Amount of patients experiencing reinfection in S-OPAT treatment | 30 days after discharge
  To investigate the amount of patients that experience reinfection when treated in S-OPAT setting
Clinical outcomes: Duration of treatment in S-OPAT | 30 days after discharge
  To investigate the amount of time patients spend in S-OPAT treatment
Clinical outcomes: Patient mortality as performing S-OPAT | 30 days after discharge
  To investigate how many patients die whilst performing S-OPAT
Adverse events | 30 days after discharge
  To investigate the adverse events reported during the first 30 days after discharge.
Readmission rate | 30 days after discharge
  To investigate the 30 day all-cause readmission rate after the end of the S-OPAT trajectory.
  To investigate the 30 day OPAT/infection related readmission rate of the S-OPAT trajectory
Satisfaction outcomes | 30 days after discharge
  To investigate the patient acceptability with S-OPAT by handing them a questionnaire about their experience with S-OPAT.
Health outcomes | 30 days after discharge
  The patients will fill out a EQ-5D-5L questionnaire both at discharge and after 30 days of S-OPAT treatment. These will be compared to each other and to other patients.

OTHER OUTCOMES:
Duration of training | 30 days after discharge
  Duration of S-OPAT training
Patient satisfaction with training | 30 days after discharge
  The patients or caregivers who followed the S-OPAT training will receive a questionnaire with questions about their experience with the training and how well they understood the training.
Difference between S-OPAT carried out by patient or caregiver | 30 days after discharge
  The performance of self-administration in the S-OPAT services by patients and caregivers will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda de Winter, PharmD, Principal Investigator — Erasmus MC University Medical Centre
Locations (2):
- Netherlands (2):
  - Amphia hospital, Breda, North Brabant
  - Erasmus MC, Rotterdam, South Holland